CLINICAL TRIAL: NCT02556476
Title: Cost Effectiveness of Intensive Care in a Low Resource Setting: Prospective Cohort of Medical Critically Ill Patients
Brief Title: Cost Effectiveness Analysis of Critical Care in Resource Limited Setting
Acronym: CEACCLR
Status: Completed | Type: Observational
Sponsor: University of Sarajevo (Other)
Responsible Party: Principal Investigator, Hajrunisa Cubro, MD, University of Sarajevo
Other Study IDs: CCUS-2435/11
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Critical Illness
Keywords: critical care; intensive care; health related quality of life; cost benefit analysis
MeSH Terms: conditions — Critical Illness | interventions — Respiration, Artificial; Ventilators, Mechanical; Neuromuscular Blockade; Renal Replacement Therapy; Hemodiafiltration; Noninvasive Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: The actual cohort of 148 critically ill medical patients that received the treatment in the intensive care unit (ICU). The interventions include interventions that are usually performed within the ICU such as mechanical ventilation, non-invasive ventilation, neuromuscular blockade, renal replacement therapy.
  Interventions: Procedure: mechanical ventilation; Procedure: neuromuscular blockade; Procedure: renal replacement therapy; Procedure: non-invasive ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — ventilator support for the patients presenting with acute respiratory failure
  Other Names: ventilator
Procedure: neuromuscular blockade — paralysis of the skeletal muscles in order to optimize mechanical ventilation, especially during ARDS
  Other Names: neuromuscular block
Procedure: renal replacement therapy — the procedures used to treat acute kidney injury
  Other Names: continuous hemofiltration (CHF) or hemodiafiltration (CHDF)
Procedure: non-invasive ventilation — Procedure used for ventilation support in patients with congestive heart failure, pulmonary edema, COPD and some other conditions.
  Other Names: continuous positive airway pressure (CPAP)

SUMMARY:
The purpose of this study was to examine the cost effectiveness of critical care in a middle income country with limited resources.

The main study hypothesis was that critical care is cost effective in low resources setting.

DETAILED DESCRIPTION:
The investigators objective was to calculate the cost effectiveness of treatment of critically ill patients in a medical ICU of a middle income country with limited access to ICU resources.

Methods: Consecutive critically ill medical patients treated in a recently established medical ICU in Sarajevo, Bosnia and Herzegovina, were prospectively recorded and a subsequent cost utility analysis of intensive care in comparison to hospital ward treatment from the perspective of health care system was performed. Incremental cost effectiveness was calculated using estimates of ICU versus non-ICU treatment effectiveness based on a formal systematic review of published studies. Decision analytic modeling was used to compare treatment alternatives. Sensitivity analyses of the key model parameters were performed.

ELIGIBILITY:
Inclusion Criteria:

* patients treated between June 1 2011 and June 29 2012 in the medical ICU

Exclusion Criteria:

* Patients who stayed in the ICU less than 24 hours and
* hospital readmissions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive critically ill patients treated during one year in a recently established medical ICU at the Sarajevo University Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
survival | one year after hospital release
  mortality was recorded one year after hospital discharge and subtracted from the value od 100% in order to get one year survival

SECONDARY OUTCOMES:
mortality | 30 days and 60 days after critical illness onset and one year after hospital release
health related quality of life (HRQOL) | one year after hospital release
  HRQOL was assessed using EQ5D-3L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hajrunisa Cubro, MD, Principal Investigator — Medical ICU University of Sarajevo Clinical Center, Sarajevo, Bosnia and Herzegovina; Ognjen Gajic, MD, MSc, Study Chair — Division of Pulmonary and Critical Care Mayo Clinic Rochester MN USA